CLINICAL TRIAL: NCT02652897
Title: Prospective Study on Hemostasis Alterations in Patients Undergoing Neuro Surgical Glioma Resection Acronym: (ABCD Study: Acute Brain Coagulopathy Development Study)
Brief Title: Hemostasis Alterations in Neurosurgical Patients
Acronym: ABCD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Santiago R. Leal-Noval (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Santiago R. Leal-Noval, Santiago R. Leal-Noval, MD, PhD, Critical Care specialist, Hospitales Universitarios Virgen del Rocío
Organization: Hospitales Universitarios Virgen del Rocío (Other)
Other Study IDs: FIS PI15 / 00512
Record Dates: First submitted 2015-12-18; First posted 2016-01-12 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Glioma; Coagulopathy; Acquired Platelet Function Disorder; Thromboelastometry; Surgery
Keywords: bleeding; clotting tests; neurosurgery; clotting time; maximum clot firmness; kinetics; lysis; primary hemostasis; platelet dysfunction; coagulation
MeSH Terms: conditions — Glioma; Hemostatic Disorders; Hemorrhage; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Exposure to glioma resection surgery: Patients undergoing elective glioma resection
  Interventions: Procedure: Exposure to glioma resection surgery
- Exposure to colon resection surgery: Patients undergoing elective colon cancer resection
  Interventions: Procedure: Exposure to colon resection surgery

INTERVENTIONS:
Procedure: Exposure to glioma resection surgery — The following blood samples will be drawn for hemostasis evaluation: 1. Conventional clotting tests, 2. Rotational thromboelastometry (ROTEM), including EXTEM and FIBTEM; 3. Platelet function as assessed by PFA-200 for; and 4. Platelet function as assessed by ara-tem, adp-tem and trap-tem. All the analyses will be performed before (within a period 24-h before surgery) and after (within of the following periods: 2 h, 24 h and 48 h after surgery).
  Groups: Exposure to glioma resection surgery
Procedure: Exposure to colon resection surgery — The following blood samples will be drawn for hemostasis evaluation: 1. Conventional clotting tests, 2. Rotational thromboelastometry (ROTEM), including EXTEM and FIBTEM; 3. Platelet function as assessed by PFA-200 for; and 4. Platelet function as assessed by ara-tem, adp-tem and trap-tem. All the analyses will be performed before (within a period 24-h before surgery) and after (within of the following periods: 2 h, 24 h and 48 h after surgery).
  Groups: Exposure to colon resection surgery

SUMMARY:
Prospective, observational study aimed to investigate the specific hemostatic alterations in patients undergoing glial tumor resection.

DETAILED DESCRIPTION:
Brain parenchyma express tissue factor and other coagulation factors in high concentrations. In addition, neuro critical patients (NCP) may present platelet dysfunction, hyperfibrinolysis, hypo coagulation and / or hyper coagulation status, early after the injury. It is not known whether these alterations of hemostasis are due to a specific brain response to aggression, or they are included into a systemic response. This prospective, observational study is aimed to investigate the coagulation disorders specifically associated with cerebral aggression.

This is a prospective, cohort study including (calculated sample size) a study group of patients undergoing elective surgery (glial tumors) and other one undergoing colo rectal surgery. Alterations of the hemostasis will be evaluated by clotting tests, thromboelastometry and tests for platelet function. Samples will be drawn before and after surgical procedures. Multiple statistical comparisons intra and inter groups will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective surgeries: glioma or colon cancer resections.

Exclusion Criteria:

* Severe bleeding leading to patient's' death.
* Incomplete tumor resection.
* Peri operative complications leading to severe bleeding or prolonged ICU or hospital stay.
* Peri operative blood components transfusion.
* Peri operative transfusion of concentrate coagulation factors.
* Intake of anti coagulant and / or antiaggregant drugs 7 days before surgery.
* History of coagulopathy.
* Inform consent denied for patients or relatives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing elective glioma (study group) and colon (control group) surgeries.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-02 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Change of INR: International Normalized Ratio | From 24-hour before surgery (baseline) at 48-hour after surgery
  Blood samples for assessing INR (clotting tests) will be drawn in these periods of time "t": "t0" (before surgery) and t1 (2-hour after surgery), t2 (24-hour after surgery) and t3 (48-hour after surgery). Changes from t0 to t1, t2 and / or t3 will be considered.
Change of aPTT: activated partial thromboplastin time (seconds). | From 24-hour before surgery (baseline) at 48-hour after surgery
  Blood samples for assessing aPTT (clotting tests) will be drawn in these periods of time "t": "t0" (before surgery) and t1 (2-hour after surgery), t2 (24-hour after surgery) and t3 (48-hour after surgery). Changes from t0 to t1, t2 and / or t3 will be considered.
Change of CT / EXTEM: clotting time (seconds). | From 24-hour before surgery (baseline) at 48-hour after surgery
  Blood samples for assessing CT / EXTEM (measured by thromboelastometry test) will be drawn in these periods of time "t": "t0" (before surgery) and t1 (2-hour after surgery), t2 (24-hour after surgery) and t3 (48-hour after surgery). Changes from t0 to t1, t2 and / or t3 will be considered.
Change of MCF / EXTEM: maximum clot firmness (mm) | From 24-hour before surgery (baseline) at 48-hour after surgery
  Blood samples for assessing MCF / EXTEM (measured by thromboelastometry test) will be drawn in these periods of time "t": "t0" (before surgery) and t1 (2-hour after surgery), t2 (24-hour after surgery) and t3 (48-hour after surgery). Changes from t0 to t1, t2 and / or t3 will be considered.
Change of ML / EXTEM: Maximum lysis (%) percentage of clot which has actually lysed | From 24-hour before surgery (baseline) at 48-hour after surgery
  Blood samples for assessing ML (measured by thromboelastometry test) will be drawn in these periods of time "t": "t0" (before surgery) and t1 (2-hour after surgery), t2 (24-hour after surgery) and t3 (48-hour after surgery). Changes from t0 to t1, t2 and / or t3 will be considered.
Change of col EPI (PFA-200): collage epinephrine bitartrate ( seconds) | From 24-hour before surgery (baseline) at 48-hour after surgery
  Blood samples for assessing col EPI (measured by platelet function analyzer : PFA-200 test) will be drawn in these periods of time "t": "t0" (before surgery) and t1 (2-hour after surgery), t2 (24-hour after surgery) and t3 (48-hour after surgery). Changes from t0 to t1, t2 and / or t3 will be considered.
Change of ara-tem / ROTEM values : platelet activation with arachidonic acid (ohm) | From 24-hour before surgery (baseline) at 48-hour after surgery
  Blood samples for assessing A6 (amplitude at 6 minutes, ohm), MS (maximum slope, ohm/min), and AUC (area under curve, ohm* min), all of then measured by platelet function analyzer ROTEM will be drawn in these periods of time "t": "t0" (before surgery) and t1 (2-hour after surgery), t2 (24-hour after surgery) and t3 (48-hour after surgery). Changes from t0 to t1, t2 and / or t3 will be considered.
Change of adp-tem / ROTEM values : platelet activation with adenosine diphosphate (ohm) | From 24-hour before surgery (baseline) at 48-hour after surgery
  Blood samples for assessing A6 (amplitude at 6 minutes, ohm), MS (maximum slope, ohm/min), and AUC (area under curve, ohm* min), all of then measured by platelet function analyzer ROTEM will be drawn in these periods of time "t": "t0" (before surgery) and t1 (2-hour after surgery), t2 (24-hour after surgery) and t3 (48-hour after surgery). Changes from t0 to t1, t2 and / or t3 will be considered.
Change of trap-tem / ROTEM values : platelet activation with thrombin activating peptide (ohm) | From 24-hour before surgery (baseline) at 48-hour after surgery
  Blood samples for assessing A6 (amplitude at 6 minutes, ohm), MS (maximum slope, ohm/min), and AUC (area under curve, ohm* min), all of then measured by platelet function analyzer ROTEM will be drawn in these periods of time "t": "t0" (before surgery) and t1 (2-hour after surgery), t2 (24-hour after surgery) and t3 (48-hour after surgery). Changes from t0 to t1, t2 and / or t3 will be considered.
Change of CT / FIBTEM: clotting time (seconds). | From 24-hour before surgery (baseline) at 48-hour after surgery
  Blood samples for assessing CT / FIBTEM (measured by thromboelastometry test) will be drawn in these periods of time "t": "t0" (before surgery) and t1 (2-hour after surgery), t2 (24-hour after surgery) and t3 (48-hour after surgery). Changes from t0 to t1, t2 and / or t3 will be considered.
Change of MCF / FIBTEM: maximum clot firmness (mm) | From 24-hour before surgery (baseline) at 48-hour after surgery
  Blood samples for assessing MCF / FIBTEM (measured by thromboelastometry test) will be drawn in these periods of time "t": "t0" (before surgery) and t1 (2-hour after surgery), t2 (24-hour after surgery) and t3 (48-hour after surgery). Changes from t0 to t1, t2 and / or t3 will be considered.
Change of coagulation factor XIII activity | From 24-hour before surgery (baseline) at 48-hour after surgery
  Factor XIII chromogenic activity assay.

SECONDARY OUTCOMES:
perioperative bleeding | from surgery to hospital discharge, an average of 2 weeks.
  Any bleeding occurring during this period.
number of days | from surgery to hospital discharge, an average of 2 weeks.
  length of stay at ICU and hospital

CONTACTS AND LOCATIONS:
Overall Officials: Santiago R. Leal-Noval, MD Ph.D, Principal Investigator — University Hospital "Virgen del Rocío", Seville, Spain
Locations (1):
- Santiago R. Leal-Noval, Seville, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leal-Noval SR, Cuenca DX, Diaz A, Fernandez-Pacheco J, Garcia-Garmendia JL, Casado M. Whole Blood Platelet Aggregation Assessed by ROTEM Platelet Equipment in Healthy Volunteers from Southern Europe: A Verification Study. J Appl Lab Med. 2023 May 4;8(3):551-558. doi: 10.1093/jalm/jfad008. PMID 36945200
- [Derived] Leal-Noval SR, Fernandez-Pacheco J, Casado-Mendez M, Cancela P, Narros JL, Arellano-Orden V, Dusseck R, Diaz-Martin A, Munoz-Gomez M. A prospective study on the correlation between thromboelastometry and standard laboratory tests - influence of type of surgery and perioperative sampling times. Scand J Clin Lab Invest. 2020 May;80(3):179-184. doi: 10.1080/00365513.2019.1704051. Epub 2019 Dec 17. PMID 31846350